CLINICAL TRIAL: NCT01940224
Title: Effectiveness of Preemptive Use of Pregabalin on Pain Intensity and Postoperative Morphine Consumption After Laparoscopic Colorectal Surgery
Brief Title: Evaluation of Preoperative Use of Pregabalin on Postoperative Analgesia After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Theodorou, MD, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UTH2828/26/06/2013
Record Dates: First submitted 2013-08-30; First posted 2013-09-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain
Keywords: Pregabalin; Laparoscopic colorectal surgery; Postoperative pain; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin & Morphine (Active Comparator): Administration of pregabalin 300 mg to patients undergo laparoscopic colorectal surgery.Patients receive oral Pregabalin 150 mg the night before surgery, and another one dose of 150 mg 1 hour prior to surgery. Postoperative administration of morphine via PCA pump for 48 hours
  Interventions: Drug: Pregabalin; Drug: Morphine
- Placebo & Morphine (Placebo Comparator): Administration of placebo to patients undergo laparoscopic colorectal surgery.Patients receive oral Placebo the night before surgery, and another one dose 1 hour prior to surgery.Postoperative administration of morphine via PCA pump for 48 hours
  Interventions: Drug: Placebo; Drug: Morphine

INTERVENTIONS:
Drug: Pregabalin — Preoperative administration of pregabalin 300mg
  Other Names: Lyrica
  Arms: Pregabalin & Morphine
Drug: Placebo — Preoperative administration of placebo
  Arms: Placebo & Morphine
Drug: Morphine — Postoperative administration of morphine via PCA pump for 48h

SUMMARY:
The purpose of this study is to evaluate how effective is the preoperative administration of pregabalin 300mg, to attenuate postoperative pain and opioids consumption after laparoscopic colorectal surgery

DETAILED DESCRIPTION:
Laparoscopic colorectal surgery has gained wide acceptance because it is associated with reduced pain, lower morbidity, faster recovery and a shorter hospital stay. However, the optimal postoperative pain management method for patients undergoing laparoscopic colorectal surgery is still under evaluation and most of the recommendations are based on studies performed in open approach procedures.

Recently, the analgesic effect of pregabalin, as a part of a multimodal analgesia, has been evaluated in many studies. They have shown that pregabalin may have a role in the post operative pain management, as an adjunct. Pregabalin is an anticonvulsant and anxiolytic drug, which have a more favorable pharmacokinetic profile from its predecessor gabapentin.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Patients who undergo laparoscopic colectomy for benign or malignant colorectal disease ( <Τ3 or =T3 tumors without distant metastasis )

Exclusion Criteria:

* Contraindication for pneumoperitoneum
* Contraindication for laparoscopic approach
* Renal or hepatic insufficiency
* Alcohol or drugs abuse
* History of chronic pain or daily intake of analgesics
* Psychiatric disorders
* Inability of patients to use PCA pump History of intake of non-steroidal anti-inflammatory drugs the last 24 hours before surgery,use of drainage after the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 48 hours
  The total dose of morphine was calculated as mg and administered by PCA pump. Postoperative morphine requirements were assessed on the arrival of the patient to the recovery room (0hrs),8 hrs,24 hrs until the completion of 48 hours after operation.

SECONDARY OUTCOMES:
Postoperative pain | 48 hours
  NRS = numeric rating scale 0-10 mm (0=no pain to 10= worst imaginable pain)
Side- effects | 48 hours
  To determine the occurrence of side effects such as postoperative nausea,vomiting, itching, headache, dizziness, blurred vision, lack of concentration, shoulder pain, sedation, and respiratory depression
Hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Elena Theodorou, MD, Principal Investigator — University Hospital of Larissa; George Tzovaras, MD, PhD, Study Chair — University Hospital of Larissa; Georgia Stamatiou, MD, PhD, Study Director — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece